CLINICAL TRIAL: NCT01396551
Title: Evaluating an Anchored Transponder in Lung Cancer Patients Receiving Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CMT - 01-10
Record Dates: First submitted 2011-07-12; First posted 2011-07-19 (Estimated); Results first posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Lung Cancer
Keywords: Anchored Beacon Transponder; Anchored Transponder; Lung cancer; Calypso system; Realtime tracking
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transponder implantation (Experimental): Implantation of anchored Beacon transponder in the lung
  Interventions: Device: Implantation of anchored Beacon transponder in the lung

INTERVENTIONS:
Device: Implantation of anchored Beacon transponder in the lung — Anchored Beacon transponder has an anchoring feature to secure it in the small airways of the lung.

SUMMARY:
Clinical study investigating the feasibility and safety of using an anchored Calypso transponder in the airways of the lung for real-time monitoring of tumor location during radiotherapy

DETAILED DESCRIPTION:
The Calypso anchored lung transponders are a modified version of the previously FDA-cleared Calypso soft tissue transponders. This modification includes an anchoring mechanism to hold the transponder positionally stable within small airways of the lung. Transponders are placed locally to the tumor within the lung and during subsequent radiotherapy the Calypso system may be used to monitor the location of the transponders and, by extension, the tumor, in real-time. This allows for improved tumor-targeting as well as gating of the radiation beam when the tumor moves outside the target field during respiratory motion.

The goals of this investigation are to show that patients with implanted anchored transponders can be localized with the Calypso System, that anchored transponder implantation and use are feasible and safe, and that anchored transponders are positionally stable in the small airways of patients with cancer of the lung.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of consent (19 years if required by local or state laws)
* Patients planning to undergo radiation therapy for primary or recurrent carcinomas of the lung or cancer that is metastatic to the lung.
* Patients who are to receive 30 Gy or more of external beam radiation therapy.
* Patients who are able to tolerate flexible bronchoscopy.
* Patients with life expectancy of at least 12 months and who are expected to be able to complete the full follow-up assessment in the protocol.
* Patients for whom the physician is able to identify suitable implantation sites for the anchored transponders on a recent (within the past 8 weeks) CT scan. This will require acquisition of a CT scan if a suitable one is not already available.
* Patients who are able to comply with the protocol.

Exclusion Criteria:

* Patients with implants in the chest region that contain metal or conductive materials (e.g., metal implants, rods, or plates) which the Sponsor considers will interfere with the Calypso System's electromagnetic localization (note that the Sponsor will review a patient's implanted metal on a case by case basis).
* Patients with active implanted devices, such as pacemakers, defibrillators, and drug infusion pumps since the effect of the Calypso System operation on these devices is unknown.
* Patients with active infections.
* Patients with bronchiectasis in the lobe of the intended implantation sites.
* Patients with a history of hypersensitivity to nickel.
* Patients whose lung tumors are being monitored with MR imaging (MR imaging of the anchored transponders is safe but yields an image artifact around the anchored transponders).
* Patients with any other medical condition or laboratory value that would, at the discretion of the investigator, preclude the patient from participation in this clinical study.
* Patients enrolled in any other clinical studies the investigator believes to be in conflict with this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Levine, PhD, Study Director — Varian Medical Systems
Locations (10):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Radiological Associates of Sacramento, Sacramento, California
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - New York University Langone Medical Center, New York, New York
  - Cancer Treatment Centers of America (CTCA), Tulsa, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
- University of Heidelberg / Thoraxklinik / DKFZ, Heidelberg, Germany
- Stellenbosch University / Tygerberg Hospital, Cape Town, South Africa
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients meeting inclusion/exclusion criteria and enrolled in the study were implanted with anchored transponders unless the patient's status changed prior to implantation. For example, if the patient's therapeutic plan was changed to exclude radiotherapy or the patient receives chest implants that preclude them from the study.
Groups:
- Transponder Implantation: Implantation of anchored Beacon transponder in the lung: Anchored Beacon transponder has an anchoring feature to secure it in the small airways of the lung. Patients were implanted with 2-3 anchored transponders prior to radiotherapy. Transponders wereused for tumor localization during radiotherapy.
Period: Overall Study
Arm/Group | Transponder Implantation
Started | 69
Completed | 69
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients who underwent implantation
Arm/Group | Transponder Implantation
Number analyzed (Participants) | 69
Age, Continuous [Median (Full Range); unit: years] | 65 [42 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 41
  South Africa | 10
  Switzerland | 10
  Germany | 8
Tumor characteristics [Count of Participants; unit: Participants]
  Primary Lung | 55
  Recurrent/second lung primary | 3
  Metastatic to the lung | 11
Co-morbidities [Count of Participants; unit: Participants]
  COPD | 46
  other cardiac disease | 14
  other pulmonary conditions | 13
  Coronary Artery Bypass graft surgery | 5
  Congestive heart failure | 4
  Prior pneumothorax | 4
  Angioplasty or coronary artery stenting | 3
Baseline symptoms [Count of Participants; unit: Participants]
  Dyspnea | 39
  Cough | 38
  Sputum production | 24
  Wheezing | 9
  Hemoptysis | 3
Prior Thoracic Surgery [Count of Participants; unit: Participants] | 15

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Proportion of Patients Who Can be Localized by the Calypso System Using the Anchored Transponders.
Description: Whether a patient can be localized by the Calypso System using the anchored transponders will be determined during the first week (i.e., the first five fractions) of radiation therapy.
Time Frame: 1-2 weeks following implantation
Population: Two patients were not included in the analysis. One patient became ineligible for Calypso localization after receiving a pacemaker, and one patient did not undergo radiation therapy because of disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Transponder Implantation
Number analyzed (Participants) | 67
Participants | 66

2. Secondary Outcome: To Assess the Implantation Procedure of the Anchored Transponder in the Lung
Description: The implantation procedure of the anchored transponder in the lung will be assessed with respect to a number of criteria: ability to implant transponders where intended, implanting physician's satisfaction with the process, and geometric configuration of the implanted transponders.
Time Frame: 1-2 weeks following implantation
Reporting Status: Not Posted

3. Secondary Outcome: To Assess the Positional Stability of the Anchored Transponders Short Term Through the Completion of Radiotherapy and Long Term Through One Year of Follow-up.
Description: The positional stability of the anchored transponder configuration will be assessed using changes in intertransponder distance. Inter-transponder distance will be calculated from CT scans acquired at treatment planning (baseline), 2-4 subsequent follow-up CT scans acquired during radiation therapy, and 4 follow-up CT scans taking place between 10-13 months post-radiotherapy
Time Frame: 1-14 months, depending on the duration of radiotherapy and time between follow-up visits.
Reporting Status: Not Posted

4. Secondary Outcome: To Evaluate Adverse Events Associated With the Anchored Transponder and the Implantation Procedure
Description: Adverse events associated with the anchored transponder and implantation procedure from the time of implantation through the completion of the follow-up period will be recorded and assessed.
Time Frame: Time of implantation through the completion of the follow-up period of the study (0-14 months)
Reporting Status: Not Posted

5. Secondary Outcome: To Collect Target Localization and Tracking Data With the Calypso System During Radiation Treatment Sessions
Description: Target localization and tracking data will be collected with the Calypso System during radiation treatment sessions.
Time Frame: Depending on the type of radiation treatment, this will take place over the course of 1-2 weeks or 1-7 weeks
Reporting Status: Not Posted

6. Secondary Outcome: To Record Usability Data, Including User Intervention in Response to the Localization and Tracking Data During the Radiation Treatment Sessions
Description: To record usability data, including user intervention in response to the localization and tracking data (e.g., pausing the bean, patient re-alignment, etc.) during the radiation treatment sessions.
Time Frame: Depending on the type of radiation treatment, this will take place over the course of 1-2 weeks or 1-7 weeks
Reporting Status: Not Posted

7. Secondary Outcome: To Calculate the Potential Reduction in Volume and Dose of Normal Lung Irradiated When a Reduced Margin is Used for the Planning Target Volume
Description: To calculate the potential reduction in volume and dose of normal lung irradiated when routine institutional planning target volume margins are reduced to a margin of 0.5 cm circumferentially made possible by realtime localization and tracking of the tumor. This calculation will be done for a subset of the patients.
Time Frame: 1-2 weeks following implantation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of patient implantation until approximately 12 months following the completion of radiotherapy.
Arm/Group | Transponder Implantation
All-Cause Mortality (participants affected / at risk) | 17/69
Serious Adverse Events (participants affected / at risk) | 7/69
Other Adverse Events (participants affected / at risk) | 36/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transponder Implantation (N=69)
Contiguous Pneumonia (Infections and infestations) | 1 (1) — Pneumonia
lung infection with pulmonary abcess and bronchopleural fistula (Infections and infestations) | 1 (1)
consolidation on major fissure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
acute bronchopneumonia (Infections and infestations) | 1 (1)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
anethesia induced short cardiac arrest (Cardiac disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transponder Implantation (N=69)
atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
imaging evidence of post obstructive pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 (10)
anchored transponder migration outside the lung (Product Issues) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 13 (13)
chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sore throat (General disorders) | 9 (9)
sputum production (General disorders) | 3 (3)
wheezing (General disorders) | 2 (2)
post extubation bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
vomiting (General disorders) | 2 (2)
excoriations in oropharynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
fatigue (General disorders) | 4 (4)
weakness (General disorders) | 1 (1)
fever (General disorders) | 3 (3)
urinary retention (Renal and urinary disorders) | 2 (2)
dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
nausea (General disorders) | 2 (2)
throat/chest tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
headache (General disorders) | 1 (1)
dry mouth (General disorders) | 1 (1)
chills (General disorders) | 1 (1)
neck pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less